CLINICAL TRIAL: NCT06810128
Title: CLINICAL PREDICTION RULE IN PROGNOSIS OF CHRONIC MECHANICAL LOW BACK PAIN AMONG HEALTH CARE PROFESSIONS
Brief Title: Predictors For the Prognosis of CMLBP Among Healthcare Professions
Status: Completed | Type: Observational
Sponsor: Alaa shaker Mohamed Mohamed (Other)
Responsible Party: Sponsor-Investigator, Alaa shaker Mohamed Mohamed, Alaa Shaker Mohamed, Cairo University
Organization: Cairo University (Other)
Other Study IDs: Predictors For CMLBP Prognosis
Record Dates: First submitted 2024-12-07; First posted 2025-02-05 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Chronic Mechanical Low Back Pain
Keywords: CMLBP among healthcare professions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Identifying clinical predictors that anticipate the prognosis of pain intensity and level of disability of mechanical low back pain among healthcare professions.It will be hypothesized that:There will be no statistical significance correlation between the prognosis of chronic mechanical low back considering pain intensity, function disability and the independant variables.

DETAILED DESCRIPTION:
The annual incidence of CMLBP among healthcare professions has been found to be 26% with a high yearly recurrence. Chronic mechanical Low back pain is the leading cause of years lived with disability worldwide. There are individual factors that can increase the risk of pain chronicity such as biomechanical, psychological, social, environmental, lifestyle, and personal factors. Therefore the main objective of the current study will be to investigate the anticipated clinical predictors that may help the prognosis of chronic mechanical LBP among health care professions. Up to author's knowledge, no studies have been carried on to identify anticipating factors related to CMLBP among healthcare professions. Studies simply identify the factors related to chronicity, they do not however study whether the presence of 1 factor is sufficient or whether a certain mix of factor is required. Therefore, the present study will be carried on to develop more comprehensive model including connections between multiple factors, in addition to consider which factors are truly important.The study procedures were explained in detail to every patient before the assessment. All patients were informed about the purpose and nature of the study, and written consent was obtained before participation in the study.

Sample size calculation is based on power analysis using the G*power program 3.1.9 (G power program version 3.1, Heinrich-Heine-University, Düsseldorf, Germany). The sample size calculation is depended on a pilot study including 10 patients diagnosed with chronic mechanical low back pain to study multi-regression between dependent variable and independent variables. The squared multiple correlation (R2) for this pilot study = 0.140. Sample size calculation based on F tests (Linear multiple regression: Fixed model, R² deviation from zero), Type I error (α) = 0.05, power (1-β error probability) = 0.80, and Effect size f2= 0.1627907 with a total sample size for 118 participants. Considering a 10% drop out rate, the appropriate minimum sample size for this study will be 130 participants diagnosed with chronic mechanical low back pain. The sample size calculation was depended on a pilot study including 10 patients diagnosed with chronic mechanical low back pain to study multi-regression between dependent variable and independent variables . The squared multiple correlation (R2) for this pilot study = 0.140. Sample size calculation based on F tests (Linear multiple regression: Fixed model, R² deviation from zero), Type I error (α) = 0.05, power (1-β error probability) = 0.80, and Effect size f2= 0.1627907 with a total sample size for 118 participants. Considering a 10% drop out rate, the appropriate minimum sample size for this study will be 130 participants diagnosed with chronic mechanical low back pain.

Statistical Analysis:

1. Statistical analysis will be conducted using SPSS Version 15.0 statistical software package (SPSS Inc, Chicago, IL, USA) to determine whether any potential prognostic variables among health care progressions with low back pain.
2. Demographic data will be expressed as mean ± standard deviation for all continuous variables and Chi square for gender distribution between groups.
3. Prior to final analysis, data will be screened for normality assumption, homogeneity of variance, and presence of extreme scores.
4. Tests of normality including Shapiro Wilk test and Kolmogorov-Smirnov test will be used.
5. Sensitivity, specificity, and positive likelihood ratios will be calculated for each potential predictor variable. To determine the most accurate set of variables for prediction of prognosis of mechanical low back pain , potential predictor variables will be entered into a step-wise logistic regression model (p<0.05).

ELIGIBILITY:
Inclusion Criteria: Subject selection based on the following criteria:

1. One hundred and thirty male and female from health care professions (Nurses, Physiotherapist, Dentists, Surgeons, Doctors, and Technicians).
2. Diagnosed with (CMLBP) (lasting for more than 3 months).
3. Age: between 30 and 49 years .
4. Subjects are at least 3/10 pain intensity on VAS.

Exclusion Criteria:

1. If investigated individuals with specific LBP (eg, infections, fracture, traumatic injuries, cancer, major systemic diseases, or congenital diseases).(Wong et al., 2022).
2. Radiculopathy/cauda equina syndrome Segmental pain
3. paresthesia in area of pain
4. loss of strength (grade 3 or less)
5. sudden loss of bladder/ bowel function
6. perianal/perineal hypaesthesia
7. death of nerve root.(Steinmetz, 2022).

Ages: 30 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1. One hundred and thirty male and female participants aged between 30 and 49 years.
  2. Health care professions (Nurses, Physiotherapists, Dentists, Doctors, surgeons, technicians), have years of experience (at least 5 years up to more than 15 years).
  3. Participants have CMLBP for at least 3 months.
  4. Chronic mechanical Low back pain (CMLBP) will be assessed by Arabic Version visual analogue scale (VAS).
  5. Functional performance will be assessed by Arabic Version Oswestery questionnaire (ODI).
  6. Fear avoidance behavior will be assessed by Arabic Version Tampa scale (TSK).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Anticipating prognosis of pain intensity and level of disability of mechanical low back pain among health care professions by identifying clinical predictors . | 1 year
  The predictors
  1-Age2-Gender 3-BMI 4-Life style5-Duration of pain 6-Intensity of pain 7-Occupation 8-Years of experience 9-Duty/Load hours 10-ODI 11-Work related frequent position12-Fear avoidance behavior Methods: 1-pain intensity will be assessed by Arabic Version(VAS).2-functional disability will be assessed by the Arabic version of (ODI ) 3-psychological status by Arabic version of Tampa scale.4-Assessment of physical activity by six-point grade.5-weight and height scale to measure weight in(kg),Height in(m). 6-BMI:weight in(kg),height in (m) will combined to measure BMI in (kg/m²)Demographic data (age, gender, occupation) will be taken .Participants will be asked about :-Duration of pain .-Years of work experience: at least 5 years, 5-10 years, 10-15 years and more than 15 years.-Duty /Load hours -Work related frequent positions (sitting, standing, squatting, slopping,, and rotation, side bending,kneeling

CONTACTS AND LOCATIONS:
Locations (1):
- Ethical research review of faculty of physical therapy Cairo university, Cairo, Egypt